CLINICAL TRIAL: NCT05821387
Title: A Randomized, Double-Blind, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Lucid-21-302 in Healthy Volunteers Under Fed and Fasted Conditions
Brief Title: Evaluating the Safety, Tolerability, Pharmacokinetics, and Effect of Food of Lucid-21-302 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quantum Biopharma (Industry)
Collaborators: Lucid Psycheceuticals Inc. (sub of FSD Pharma, Inc.) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Lucid-21-302-001; 2786 (Other: Biopharma Services Incorporated)
Record Dates: First submitted 2023-03-21; First posted 2023-04-20 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: 5 SAD Cohorts. Each SAD cohort will enroll 8 participants randomized 6 active:2 placebo to receive single doses of Lucid-21-302. For SAD cohort with food effect, all 8 participants will receive Lucid-21-302.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lucid-21-302 (Experimental): Single-ascending dose cohorts
  Interventions: Drug: Lucid-21-302
- Placebo (Placebo Comparator): Single-ascending dose cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lucid-21-302 — A small molecule inhibitor of hypercitrullination
  Arms: Lucid-21-302
Drug: Placebo — Product containing excipients with no active ingredients
  Arms: Placebo

SUMMARY:
This study aims to determine the safety, tolerability, and pharmacokinetics of single doses of Lucid-21-302 in healthy adult volunteers. This study will also investigate the effects of food in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers, 18 - 60 years of age, inclusive at the time of informed consent.
2. Body mass index (BMI) that is within 18.5 - 30.0 kg/m2, inclusive, and minimum weight of 50 kg.
3. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
4. QTcF interval ≤ 440 msec for males and ≤ 460 msec for females, unless deemed otherwise by the PI/Sub-Investigator.
5. Systolic blood pressure between 95 - 140 mmHg, inclusive, and diastolic blood pressure between 55 - 90 mmHg, inclusive, and heart rate between 50 - 100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
6. Clinical laboratory values within the laboratory test ranges and/or values in the clinical site's SOPs that are classified as "Not Clinically Significant."
7. Non-smoker and non-nicotine user, for at least six months prior to study drug administration.
8. Ability to comprehend and be informed of the nature of the study, as assessed by PI. Capable of giving written informed consent prior to any study related procedure. Must be able to communicate effectively with clinic staff.
9. Ability to speak, read, and understand English sufficiently to allow completion of all study assessments.
10. Ability to consume standard meals and the ability to fast for at least 14 hours for the SAD study and at least ten hours for the MAD study.
11. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
12. Agree not to have a tattoo or body piercing until the end of the study.
13. Agree not to receive the COVID-19 vaccination or other vaccination from seven days prior to the study drug dose until seven days after study drug administration in the study.
14. Agree not to drive or operate heavy machinery if feeling dizzy, drowsy, or otherwise mentally impaired following study drug administration until full mental alertness is regained.
15. Female participants must be non-pregnant and non-lactating and fulfill at least one of the following:

    * Be surgically sterile for a minimum of six months (achieved through hysterectomy, oophorectomy, or bilateral salpingectomy; note that tubal ligation is not considered a method of permanent sterilization).
    * Post-menopausal for a minimum of one year (postmenopausal is confirmed by serum FSH values collected at screening).
    * Agree to avoid pregnancy and use an acceptable effective method of contraception with male sexual partners from at least 30 days prior to the study until at least 30 days after the study has ended (last study procedure).
    * Acceptable effective methods of contraception include using a male condom in conjunction with non-hormonal contraceptives, such as a non-hormonal intrauterine device; or a double-barrier method (e.g., male condom with diaphragm and spermicide used simultaneously, male condom with cervical cap and spermicide used simultaneously). Abstinence as a method of contraception is acceptable if it is in line with the preferred and usual lifestyle of the study participant.
16. Males who are able to father children must agree to use an acceptable effective method of contraception with female sexual partners of childbearing potential and not donate sperm during the study and for at least 90 days after the last dose of the study drug (Lucid-21-302 or placebo).

    * Acceptable effective methods of contraception include using a male condom with a female sexual partner of childbearing potential who is using oral contraceptives, hormonal patch, implant or injection, intrauterine device or system; or a double-barrier method (e.g., male condom with diaphragm and spermicide used simultaneously, male condom with cervical cap and spermicide used simultaneously). Abstinence as a method of contraception is acceptable if it is in line with the preferred and usual lifestyle of the study participant.
    * If a participant's partner becomes pregnant during his participation in the study and for 90 days after he has completed his last study drug administration, he must inform site staff immediately.
17. Deemed suitable for the study by the PI/Sub-Investigator and/or clinical staff.

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.

   o AST, ALP, ALT, bilirubin, and/or GGT levels that are outside of normal laboratory ranges
2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within seven days prior to first study drug administration, as determined by the PI/Sub-Investigator.
3. History of seizures, family history of seizures, history of head trauma, history of neurosurgery, or first-degree relative with idiopathic generalized epilepsy or other congenital epilepsies.
4. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
5. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
6. A positive test result for human immunodeficiency virus (HIV), chronic Hepatitis B surface antigen, or Hepatitis C.
7. A positive test result for drugs with abuse potential (cannabis, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), breath alcohol test or urine cotinine test.
8. Positive pregnancy test for female participants.
9. Known history or presence of:

   * Food allergies;
   * Presence of any dietary restrictions unless deemed by the PI/Sub-I as "Not Clinically Significant;"
   * Severe allergic reactions (e.g., anaphylactic reactions, angioedema).
10. Intolerance to and/or difficulty with blood sampling through venipuncture.
11. Individuals who have donated, in the days prior to first study drug administration:

    * 50-499 mL of blood in the previous 30 days;
    * 500 mL or more in the previous 56 days.
12. Donation of plasma by plasmapheresis within 7 days prior to study drug administration.
13. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to study drug administration.
14. Use of any enzyme-modifying drugs and/or other products, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort, and rifampicin) in the previous 30 days before study drug administration.
15. Use of any prescription medication within 14 days prior to study drug administration.
16. Use of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements) within 14 days prior to study drug administration.
17. Consumption of food or beverages containing grapefruit and/or pomelo within 10 days prior to study drug administration.
18. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hr before dosing (includes coffee and tea).
19. Individuals having undergone any major surgery within six months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.
20. Have any other conditions that, in the opinion of the Investigator or Sponsor, would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the study.
21. Difficulty with swallowing tablets or capsules.
22. Have had a tattoo or body piercing within 30 days prior to study drug administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Single Dose Safety Outcome Measures | Up to 12 days
  Incidence and severity of adverse events (AEs), laboratory, ECG, physical exam, neurological exam and vital sign changes
AUC from time zero to the last non-zero concentration after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
Cmax after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
Tmax after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
AUC0-inf after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
t1/2 after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
Kel after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
CL/F after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
Vd/F after single dose | Pre-dose to 48 hours post-dose
  PK characteristics after single dose
Effect of Food on the single dose AUC from time zero to the last non-zero concentration | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose Cmax | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose Tmax | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose AUC0-inf | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose t1/2 | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose Kel | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose CL/F | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose Vd/F | Pre-dose to 48 hours post-dose
  Effect of food on the single dose PK

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Szeto, MD, Principal Investigator — Biopharma Services Incorporated
Locations (1):
- Biopharma Services Incorporated, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tejeda EJC, Bello AM, Wasilewski E, Koebel A, Dunn S, Kotra LP. Noncovalent Protein Arginine Deiminase (PAD) Inhibitors Are Efficacious in Animal Models of Multiple Sclerosis. J Med Chem. 2017 Nov 9;60(21):8876-8887. doi: 10.1021/acs.jmedchem.7b01102. Epub 2017 Oct 30. PMID 29045782
- [Background] Caprariello AV, Rogers JA, Morgan ML, Hoghooghi V, Plemel JR, Koebel A, Tsutsui S, Dunn JF, Kotra LP, Ousman SS, Wee Yong V, Stys PK. Biochemically altered myelin triggers autoimmune demyelination. Proc Natl Acad Sci U S A. 2018 May 22;115(21):5528-5533. doi: 10.1073/pnas.1721115115. Epub 2018 May 4. PMID 29728463
- See also: Website for FSD Pharma Inc. — https://fsdpharma.com/